CLINICAL TRIAL: NCT06305390
Title: Fully Hybrid 18F-PSMA PET/MRI as One-stop Approach for the Diagnosis of Clinically Significant Prostate Cancer.
Acronym: RF2021-1237227
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Chiti Arturo, PI, IRCCS San Raffaele
Other Study IDs: 2022-003905-31
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-09

CONDITIONS: Clinical Suspicion of Prostate Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- single arm
  Interventions: Diagnostic Test: PET/MRI

INTERVENTIONS:
Diagnostic Test: PET/MRI — 18F-PSMA PET/MRI

SUMMARY:
This project aims to evaluate the role of fully hybrid PET/MRI with 18FPSMA and multiparametric MR imaging (mpMRI) as one-stop approach for the diagnosis of clinically significant prostate cancer (csPCa).

Our main hypothesis is that adding 18F-PSMA PET to mpMRI prior to biopsy, will reduce the number of false negative findings, while at the same time, allowing also to reduce the number of unnecessary prostate biopsies in patients with low-risk, clinically indolent PCa.

ELIGIBILITY:
Inclusion Criteria:

1. Men at least 18 years of age referred with clinical suspicion of prostate cancer candidate for prostate biopsy
2. Feasibility to undergo all procedures listed in protocol
3. Ability to provide written informed consent

Exclusion Criteria:

1. Prior diagnosis of prostate cancer
2. Contraindication to MRI (e.g. claustrophobia, pacemaker, estimated GFR lower or equal to 50mls/min)
3. Contraindication to prostate biopsy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with clinical suspicion of clinically significant prostate cancer (csPCa).
Sampling Method: Probability Sample
Enrollment: 167 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
To assess the accuracy and the predictive value of fully hybrid 18F-PSMA PET/MRI for the diagnosis of clinically significant prostate cancer (csPCa) | PET/MRI: day 0 prostate biopsy: day 0-90 days
  Diagnostic accuracies of 18F-PSMA PET and mpMRI will be calculated by means of sensitivity: true positive/(true positive + false negative) and specificity: true negative/(false positive + true negative) using the prostate biopsy result as reference standard.

SECONDARY OUTCOMES:
To compare the proportion of csPCa missed by 18F-PSMA PET scan or mpMRI alone To report the reduction in the detection of clinically insignificant PCa when combining mpMRI and 18F-PSMA PET | PET/MRI: day 0 prostate biopsy: day 0-90 days
  The proportion of csPCa (defined by analysis of prostate biopsy cores, ISUP grade equal or higher than 2) missed by PSMA PET scan or mpMRI alone will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Chiti, MD, Study Director — IRCCS Ospedale San Raffaele
Locations (1):
- U.O. of Nuclear Medicine, ,Ospedale San Raffaele, Milan, Italy